CLINICAL TRIAL: NCT00457470
Title: A Phase 2, Multi-Stage, Multi-Center Trial Exploring The Safety And Efficacy Of AG-014699 In Subjects With Diffuse Diabetic Macular Edema (DME) Involving The Center Of The Retina
Brief Title: A Phase 2 Study Exploring The Safety And Efficacy Of Novel Drug Treatment In Subjects With Diabetic Macular Edema (DME)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Cancelled before first patient enrolled
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4991010
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy | interventions — rucaparib

INTERVENTIONS:
Drug: AG-014699

SUMMARY:
This study will evaluate the safety and efficacy of AG-014699 in diabetic patients

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients, either man or woman, with diabetic retinopathy, at least 18 years of age

Exclusion Criteria:

* patients treated with laser therapy within the last 90 days
* patients with likelyhood to require cataract surgery within 3 months
* Uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06

PRIMARY OUTCOMES:
Change of retinal thickness at Day 15 or Day 25 depending on dosing regimen

SECONDARY OUTCOMES:
Proportion of subjects with reduction in retinal thickness from baseline in 2 months
Change in retinal thickness for 2 months
Change in visual acuity for 2 months
; Proportion of eyes experiencing an improvement in the degree of retinopathy at Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4991010&StudyName=A%20Phase%202%20Study%20Exploring%20The%20Safety%20And%20Efficacy%20Of%20Novel%20Drug%20Treatment%20In%20Subjects%20With%20Diabetic%20Macular%20Edema%20%28DME%29